CLINICAL TRIAL: NCT06057636
Title: Hypnosis for Pain in Black Women With Advanced Breast Cancer: A Feasibility Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit participants
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: Baylor University (Other)
Responsible Party: Principal Investigator, Noel Arring, Associate Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UTK-IRB-23-07650-XP
Record Dates: First submitted 2023-09-19; First posted 2023-09-28 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Inflammatory Breast Cancer Stage IV; Inflammatory Breast Neoplasms; Triple Negative Breast Neoplasms; Neoplasm Metastasis
Keywords: breast cancer; cancer pain; pain management; hypnosis; Black or African American
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms; Triple Negative Breast Neoplasms; Neoplasm Metastasis; Cancer Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: This is a two-arm, randomized clinical trial.
Who Masked: Participant
Masking Description: single-masking, participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Administered Hypnosis (Experimental): Self-administered hypnosis will be practiced daily, at home for 6 weeks. Hypnosis sessions are expected to last ~20 minutes. Practices using the recordings will be documented on the Hypnosis Practice Log.
  Interventions: Behavioral: Self-Administered Hypnosis
- Self Administered White Noise Hypnosis (Active Comparator): Self-administered white noise hypnosis will be practiced daily using a white noise recording. Participants will practice hypnosis at home after completing the virtual consent/baseline visit and the virtual education visit.
  Interventions: Behavioral: Self-Administered White Noise Hypnosis

INTERVENTIONS:
Behavioral: Self-Administered Hypnosis — Participants will choose from one of three 20-minute prerecorded hypnosis audio files. Practices using the recordings will be documented on the hypnosis practice log.
  Arms: Self-Administered Hypnosis
Behavioral: Self-Administered White Noise Hypnosis — Participants will be listening to the same 20-minute white noise audio recording for 6 weeks and will be encouraged to practice daily. Practices using the recordings will be documented on the hypnosis practice log.
  Arms: Self Administered White Noise Hypnosis

SUMMARY:
The purpose of this study is to compare two hypnotic interventions for Black women with advanced cancer pain in preparation for a well-powered phase III study. The investigators plan to enroll 30 adult Black women with advanced cancer pain in a 2-arm pilot randomized controlled trial (RCT).

The primary aim will be to evaluate the feasibility of conducting the 2-arm clinical trial. It is hypothesized that at least 75% of participants in both study arms will complete study requirements. The secondary aims will be to evaluate the participant's experience with the intervention and to determine the effect size of the intervention on pain severity.

DETAILED DESCRIPTION:
Envision is a randomized, 2-arm, mixed-methods pilot study to evaluate the feasibility of translating a promising in-person hypnosis intervention for advanced cancer pain into a culturally appropriate, remotely delivered hypnosis intervention for pain in Black women with advanced cancer. The study is 6 weeks long and does not require any in-person visits. If a breast cancer survivor is determined eligible, they will be educated on the purpose, requirements, and procedures. If interested, participants will be emailed the consent form and will schedule a virtual consent/baseline visit. After consent is obtained, the participant will be randomly assigned to one of two types of hypnotic relaxation to be used alongside current pain treatment using 1:1 randomization and given a study number. The participant will complete online surveys at the virtual baseline visit. An MP3 player with hypnotic relaxation audio files will be sent to the participant's address and a virtual education visit will be scheduled. At this second virtual visit, participants will receive education about their study arm and a start date will be agreed upon for week 1. Beginning week 1 and continuing through week 6, participants will listen to their assigned hypnotic relaxation audio files daily and be asked to complete a weekly practice log. Participants will also continue to meet with study staff virtually for weekly check-ins. At these weekly meetings, progress and adverse events will be assessed and relevant online surveys will be completed.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older Black female
2. Diagnosed with Stage IV Breast Cancer with life expectancy of 6 months or more
3. Ability to read and write English
4. Ability to complete questionnaire(s) by themselves or with assistance.
5. Report cancer-related pain that they rate as ≥4 on a numeric pain rating scale of 0-10 with 0 being "no pain" and 10 being "the worst it can be" for the past month or more.
6. Ability to provide informed written consent.

Exclusion Criteria:

1. Diagnosis of major depressive disorder or acute anxiety disorder per the medical record or self-report in the past 2 years
2. Serious psychological illness, specifically psychoses, schizophrenia, or borderline personality disorder per the medical record or self-report
3. Currently enrolled in hospice
4. Currently using hypnosis for any reason
5. Non-English speaking
6. Unable to complete questionnaires or follow directions independently.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Screen failure rate (a measure of feasibility) | Recruitment to screening (up to 3 months)
  The number of women screened ineligible
Accrual rate (a measure of feasibility) | Screening to consent (up to 30 days)
  The number of participants who consented divided by the number eligible
Retention rate / acceptability (a measure of feasibility) | Baseline through study completion, 6 weeks
  The number of participants who complete the 6 weeks of the study divided by the number who consented.

SECONDARY OUTCOMES:
Participant experience | consent to week 6
  Determine factors affecting participant experience through open-ended interview questions.
Pain severity and Interference | consent to week 6
  Change in Brief Pain Inventory-Short Form scores. The Brief Pain Inventory-Short Form contains two subscales, pain severity and pain interference. Both scales include individual items that are scored on a scale of 0-10. The pain severity scale includes 4 items, with a possible range of 0-40. The pain interference scale includes 7 items, with a possible range 0-70. Higher scores indicate greater pain severity and greater pain interference.

CONTACTS AND LOCATIONS:
Overall Officials: Noel M Arring, DNP, PhD, RN, Principal Investigator — University of Tennessee Knoxville
Locations (1):
- University of Tennessee Knoxville, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
This is a small pilot study and as such, data will be thoroughly interrogated. However, if an investigator feels there are unanswered questions or wishes to add to a larger dataset, we would entertain all data-sharing requests for deidentified data as appropriate.